CLINICAL TRIAL: NCT00644358
Title: A One Year Open Label Study Assessing the Safety and Tolerability of Vilazodone in Patients With Major Depressive Disorder
Brief Title: A One Year Open Label Study Assessing the Safety and Tolerability of Vilazodone in Patients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDA-07-DP-04
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vilazodone (Experimental): Vilazodone titrated up to 40 mg/day for 1 year.
  Interventions: Drug: vilazodone

INTERVENTIONS:
Drug: vilazodone — titration to 40 milligrams (mg) every day (qd) for 1 year
  Other Names: EMD 68843, SB-659746

SUMMARY:
This open label 52-week clinical trial is designed to assess the safety and tolerability of vilazodone and to analyze genetic markers of response to vilazodone in adult patients diagnosed with MDD. This study will enroll approximately 600 patients.

DETAILED DESCRIPTION:
Patients will be enrolled at approximately 40 US investigative sites and receive vilazodone for 52 weeks of open label treatment. Safety measurements will include adverse events, vital signs, laboratory, ophthalmologic exams, Changes in Sexual Function Questionnaire (CSFQ) scale and electrocardiogram (ECG) findings collected over the course of the treatment period. Effectiveness measurements will be done at baseline and each visit until week 52 or end-of-treatment. A deoxyribonucleic acid (DNA) sample will be collected for genetic analysis related to response to vilazodone.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18-70 years of age.
* Meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder.
* Hamilton Depression Rating Scale (HAM-D) score ≥ 18 on the first 17 items of the 21-item HAM-D at Screening and Baseline Visits.
* Patients must have general ocular health.

Exclusion Criteria:

* Patients with a history of schizophrenia, schizoaffective disorder or bipolar I or II disorder (with a history of hypomanic or manic episodes).
* Patients who meet DSM-IV-TR criteria for substance abuse or dependence within 1 year of the Baseline visit.
* Patients who, in the Investigator's judgment, pose a serious suicidal or homicidal risk or have made a suicide attempt within 6 months prior to Screening Visit.
* Patients who are taking psychotropic drugs. Patients who have taken psychotropic drugs must have discontinued these prior to Screening Visit.
* Patients taking migraine medications with a serotonergic mechanism of action.
* Patients taking Cytochrome P450 3A4 (CYP3A4) inhibitors such as grapefruit juice, ketoconazole, diltiazem, and macrolide antibiotics.
* Patients with a known hypersensitivity to selective serotonin reuptake inhibitors (SSRIs) or 5-hydroxytryptamine 1a (5-HT1a) agonists.
* Patients previously treated with vilazodone.
* Patients taking Chantix or St. John's Wort.
* Presence of significant acute or chronic medical disorders by history or physical exam.
* Patients with a history of seizure disorders.
* Prior history of malignancy if patient has <5 year survival OR completed treatment <1 year prior to enrollment and is currently without evidence of recurrence.
* Skin cancers other than malignant melanoma will be permitted.
* Patients with evidence of other central nervous system disorders including psychosis, delirium, dementia and amnesic disorders.
* Patients with renal impairment or hepatic impairment.
* Patients who are not euthyroid.
* Patients with any serious medical or neurological disorder or condition that make it unlikely that the patient could complete one year of treatment or would otherwise preclude the administration of study medication.
* Female patients must not be pregnant, not lactating, and not planning to become pregnant during the time of study participation. All female patients who are not at least 1 year post menopausal or irreversibly surgically sterilized must be using adequate and reliable contraception throughout the trial.
* Patients with clinically significant ECG abnormalities which, as determined by the investigator, make it unlikely that the patient would complete one year of treatment or would otherwise preclude treatment with vilazodone.
* Patients having clinically significant abnormal laboratory findings.
* Patients with a positive drug screen.
* Patients who, in the opinion of the investigator, would be noncompliant with the visit schedule or study procedures.
* Patients that have taken an investigational drug or participated in an investigational drug trial within the past 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2007-12-31 (Actual); Primary Completion 2009-05-31 (Actual); Study Completion 2009-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol R Reed, MD, Study Director — Forest Laboratories
Locations (38):
- United States (38):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Affiliated Research Institute, San Diego, California
  - Collaborative Neuroscience Network, Inc, Torrance, California
  - Pacific Clinical Research, Upland, California
  - Radiant Research, Denver, Colorado
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Lady Lake, Florida
  - Clinical Neuroscience Solutions, PA, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Carman Research, Smyrna, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Davis Clinic, Indianapolis, Indiana
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Capital Clinical Research Associates, Rockville, Maryland
  - Summit Research Network, Farmington, Michigan
  - Radiant Research, St Louis, Missouri
  - Radiant Research, Las Vegas, Nevada
  - Bioscience Research, LLC, Mount Kisco, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - North Coast Clinical Trials, Beachwood, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Introspect of Buxmont, Colmar, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - FutureSearch Trials, Dallas, Texas
  - Croft Group Research Center, San Antonio, Texas
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Neuroscience, Inc., Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia

REFERENCES:
- [Derived] Jain R, Chen D, Edwards J, Mathews M. Early and sustained improvement with vilazodone in adult patients with major depressive disorder: post hoc analyses of two phase III trials. Curr Med Res Opin. 2014 Feb;30(2):263-70. doi: 10.1185/03007995.2013.855188. Epub 2013 Oct 31. PMID 24127687
- [Derived] Clayton AH, Kennedy SH, Edwards JB, Gallipoli S, Reed CR. The effect of vilazodone on sexual function during the treatment of major depressive disorder. J Sex Med. 2013 Oct;10(10):2465-76. doi: 10.1111/jsm.12004. Epub 2012 Dec 6. PMID 23216998
- [Derived] Reed CR, Kajdasz DK, Whalen H, Athanasiou MC, Gallipoli S, Thase ME. The efficacy profile of vilazodone, a novel antidepressant for the treatment of major depressive disorder. Curr Med Res Opin. 2012 Jan;28(1):27-39. doi: 10.1185/03007995.2011.628303. Epub 2011 Nov 23. PMID 22106941
- [Derived] Robinson DS, Kajdasz DK, Gallipoli S, Whalen H, Wamil A, Reed CR. A 1-year, open-label study assessing the safety and tolerability of vilazodone in patients with major depressive disorder. J Clin Psychopharmacol. 2011 Oct;31(5):643-6. doi: 10.1097/JCP.0b013e31822c6741. PMID 21869687

RESULTS

PARTICIPANT FLOW:
Groups:
- Vilazodone: Vilazodone titrated up to 40 milligrams (mg)/day for 1 year.
Period: Overall Study
Arm/Group | Vilazodone
Started | 616
Completed | 254
Not Completed | 362
Not completed — Adverse Event | 124
Not completed — Lost to Follow-up | 105
Not completed — Consent Withdrawal | 64
Not completed — Lack of Effectiveness | 39
Not completed — Protocol Violation | 5
Not completed — Noncompliance | 14
Not completed — Other Unspecified | 11

BASELINE CHARACTERISTICS:
Population: Safety population consisted of enrolled participants who took at least 1 dose of study drug and had at least 1 post-baseline safety measurement.
Arm/Group | Vilazodone
Number analyzed (Participants) | 599
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 407
  Male | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 545
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 103
  White | 479
  More than one race | 0
  Unknown or Not Reported | 1
Height [Mean (Standard Deviation); unit: cm] | 168.4 (9.62)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant administered study drug. An AE could, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not related to the medicinal product. An AE that occurred during the treatment period was defined as a TEAE if the AE was either not present at, or before, the day of the first dose of study medication or was present at, or before, the day of the first dose of study medication and increased in severity during the treatment period. AEs included abnormal clinically significant findings for laboratory parameters, physical examinations, vital signs, weight, electrocardiograms (ECGs), the Change in Sexual Functioning Questionnaire (CSFQ), ophthalmologic exams and the Columbia-Suicide Severity Rating Scale (C-SSRS).
Time Frame: From first dose of study medication and up to 30 days after the last dose of study medication (Up to 13 months)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Vilazodone
Number analyzed (Participants) | 599
Participants | 562

2. Secondary Outcome: Change Form Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a clinician-rated scale for assessing depressive symptomatology that had occurred in participants during the week preceding each interview. Participants were rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest. Each item was scored on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score was the sum of the scores on the 10 items and ranged from 0 to 60. A higher score indicated more depressive symptomatology. A negative change score indicated improvement.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6 ,8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52/Early Termination
Population: Effectiveness Population consisted of all participants who took at least one dose, and had at least one post-baseline efficacy endpoint measurement. The number analyzed for each category row is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vilazodone
Number analyzed (Participants) | 596
score on a scale
  Baseline | 29.9 (4.45)
  Change from Baseline at Week 1 | -4.7 (5.38)
  Change from Baseline at Week 2 | -9.3 (6.72)
  Change from Baseline at Week 3 | -13.0 (7.76)
  Change from Baseline at Week 4 | -14.9 (7.99)
  Change from Baseline at Week 6 | -17.1 (8.28)
  Change from Baseline at Week 8 | -18.5 (8.38)
  Change from Baseline at Week 12 | -19.9 (8.31)
  Change from Baseline at Week 16 | -20.6 (8.31)
  Change from Baseline at Week 20 | -21.1 (8.39)
  Change from Baseline at Week 24 | -21.7 (7.81)
  Change from Baseline at Week 28 | -21.6 (7.99)
  Change from Baseline at Week 32 | -21.9 (8.26)
  Change from Baseline at Week 36 | -22.1 (7.89)
  Change from Baseline at Week 40 | -22.7 (7.33)
  Change from Baseline at Week 44 | -21.9 (8.12)
  Change from Baseline at Week 48 | -22.5 (7.92)
  Change from Baseline at Week 52 | -22.8 (7.89)
  Change from Baseline at Early Termination | -10.9 (9.78)

3. Secondary Outcome: Change From Baseline in Clinical Global Impressions - Severity (CGI-S) Score
Description: The CGI-S is a clinician-rated scale that measures global severity of illness at a given point in time using a 7-point scale where 1=normal, not at all ill, and 7=among the most severely ill. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6 ,8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52/Early Termination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vilazodone
Number analyzed (Participants) | 596
score on a scale
  Baseline | 4.3 (0.52)
  Change from Baseline at Week 1 | -0.3 (0.57)
  Change from Baseline at Week 2 | -0.7 (0.83)
  Change from Baseline at Week 3 | -1.1 (1.04)
  Change from Baseline at Week 4 | -1.4 (1.12)
  Change from Baseline at Week 6 | -1.7 (1.18)
  Change from Baseline at Week 8 | -1.9 (1.21)
  Change from Baseline at Week 12 | -2.1 (1.18)
  Change from Baseline at Week 16 | -2.3 (1.13)
  Change from Baseline at Week 20 | -2.4 (1.15)
  Change from Baseline at Week 24 | -2.4 (1.09)
  Change from Baseline at Week 28 | -2.4 (1.09)
  Change from Baseline at Week 32 | -2.5 (1.11)
  Change from Baseline at Week 36 | -2.5 (1.13)
  Change from Baseline at Week 40 | -2.5 (1.05)
  Change from Baseline at Week 44 | -2.4 (1.12)
  Change from Baseline at Week 48 | -2.5 (1.08)
  Change from Baseline at Week 52 | -2.6 (1.13)
  Change from Baseline at Early Termination | -1.0 (1.21)

4. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: The CGI-I is a clinician-rated scale for assessing improvement of a patient's condition, using a 7-point scale where 1=very much improved (best) and 7=very much worse.
Time Frame: Weeks 1, 2, 3, 4, 6 ,8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52/Early Termination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vilazodone
Number analyzed (Participants) | 596
score on a scale
  Week 1 | 3.5 (0.67)
  Week 2 | 3.0 (0.85)
  Week 3 | 2.5 (0.94)
  Week 4 | 2.3 (0.94)
  Week 6 | 2.0 (0.92)
  Week 8 | 1.9 (0.93)
  Week 12 | 1.7 (0.93)
  Week 16 | 1.6 (0.90)
  Week 20 | 1.5 (0.84)
  Week 24 | 1.5 (0.75)
  Week 28 | 1.5 (0.79)
  Week 32 | 1.5 (0.83)
  Week 36 | 1.5 (0.78)
  Week 40 | 1.4 (0.74)
  Week 44 | 1.5 (0.86)
  Week 48 | 1.4 (0.74)
  Week 52 | 1.4 (0.75)
  Early Termination | 2.9 (1.18)

ADVERSE EVENTS:
Time Frame: From first dose of study medication and up to 30 days after the last dose of study medication (Up to 13 months)
Arm/Group | Vilazodone
Serious Adverse Events (participants affected / at risk) | 23/599
Other Adverse Events (participants affected / at risk) | 497/599
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vilazodone (N=599)
Duodenal stenosis (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Bronchoscopy (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Serotonin syndrome (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Panic attack (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vilazodone (N=599)
Diarrhoea (Gastrointestinal disorders) | 214
Dry mouth (Gastrointestinal disorders) | 66
Nausea (Gastrointestinal disorders) | 189
Vomiting (Gastrointestinal disorders) | 44
Fatigue (General disorders) | 46
Nasopharyngitis (Infections and infestations) | 45
Upper respiratory tract infection (Infections and infestations) | 82
Urinary tract infection (Infections and infestations) | 35
Weight increased (Investigations) | 57
Increased appetite (Metabolism and nutrition disorders) | 54
Back pain (Musculoskeletal and connective tissue disorders) | 33
Dizziness (Nervous system disorders) | 64
Headache (Nervous system disorders) | 120
Somnolence (Nervous system disorders) | 64
Abnormal dreams (Psychiatric disorders) | 62
Anxiety (Psychiatric disorders) | 36
Insomnia (Psychiatric disorders) | 78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.